CLINICAL TRIAL: NCT05592548
Title: Open Label Split Face Pilot Study to Assess the Safety and Efficacy of Cold Atmospheric Plasma (non-thermal Plasma) for the Treatment of Rosacea
Brief Title: Rosacea Treatment Using Non-thermal (cold) Atmospheric Plasma Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Skin Center Dermatology Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROSACECAPRCM
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Rosacea, Papulopustular
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: split face study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study (Experimental): Single arm study: split face treatment
  Interventions: Device: cold atmospheric plasma

INTERVENTIONS:
Device: cold atmospheric plasma — Cold atmospheric plasma will be generated on the skin surface using an electric device

SUMMARY:
10-13 patients will be enrolled to receive split face treatment: the control side will be treated with metronidazole cream, the intervention side will be treated with a cold atmospheric plasma device

ELIGIBILITY:
Inclusion Criteria:

* Papulopustular rosacea of the cheeks
* Ability to complete six weeks of twice-weekly treatments

Exclusion Criteria:

* substantial asymmetry of disease distribution
* previous failure of topical ivermectin treatment
* presence of any other facial dermatoses
* presence of any photosensitizing disorders
* systemic tetracycline, systemic or topical ivermectin treatment within 6 weeks of start date
* current or within prior 3 months treatment with systemic immune-suppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy - Investigator global assessment | 6 weeks
  Rosacea improvement will be evaluated based on clinical photos (worsened, unchanged, mild improvement, substantial improvement, cleared)
RosaQoL change | 6 weeks
  Rosacea Quality of Life tool: 5-point scale Ranging from 1 (no impact) to 5 (worst impact)
Demodex count change | 6 weeks
  Change in demodex folliculorum mite density, measured by Reflectance Confocal Microscopy )number of follicles with mite, total number of mites in measured area, number of mites per follicle)
Efficacy - National Rosace Society Expert Committee grading system | 6 weeks
  Complex scoring system as described by Wilkin et al, J Am Acad Dermatol 2004;50:907-12

SECONDARY OUTCOMES:
Tolerability - Incidence of Treatment-Emergent Adverse Events as assessed by patient review | 6 weeks
  patient reported adverse effects collected using questionnaires
Tolerability - pain as assessed by NRS scale | 6 weeks
  Pain assessment using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

CONTACTS AND LOCATIONS:
Overall Officials: Peter Friedman, MD PhD, Principal Investigator — The Skin Center Dermatology Group
Locations (1):
- The Skin Center Dermatology Group, New City, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malik S, Gill M, Fridman G, Fridman A, Friedman PC. Cold atmospheric plasma reduces demodex count on the face comparably to topical ivermectin, as measured by reflectance confocal microscopy. Exp Dermatol. 2022 Sep;31(9):1352-1354. doi: 10.1111/exd.14584. Epub 2022 May 11. No abstract available. PMID 35491738